CLINICAL TRIAL: NCT05737732
Title: Systematic Light Exposure Effects on Circadian Rhythms Entrainment, Inflammation, Neutropenic Fever and Symptom Burden Among Multiple Myeloma Patients Undergoing Autologous Stem Cell Transplantation
Brief Title: The Ambient Light Multiple Myeloma Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Director of Light and Health Research Center at Mount Sinai, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-21-01146
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circadian Effective Lighting (CEL) (Active Comparator): The CEL will be performed in hospital sites over a 2-month period.
  Interventions: Device: Circadian Effective Lighting
- Circadian Ineffective Lighting (CIL) (Sham Comparator): The comparator lighting will be performed identical to Arm 1, at specified lower levels of lighting.
  Interventions: Device: Circadian Ineffective Lightning (CIL)

INTERVENTIONS:
Device: Circadian Effective Lighting — Participants will receive lighting with a spectrum of 300K, 500 lux to the eye level between 7:00am and 10:00am in the morning, and hospital lighting (<100lux) during the afternoon between 10:00am and 6:00pm. In the evening this group of participants will receive lighting with a spectrum of 3000K, <50lux at eye light level between 6:00PM and bedtime.
  Arms: Circadian Effective Lighting (CEL)
Device: Circadian Ineffective Lightning (CIL) — Participants will receive lower lighting levels in the morning (lighting with A spectrum of 300k, <50lux to the eye level between 7:00am and 10:00am) and the same lighting levels throughout the rest of the day.
  Arms: Circadian Ineffective Lighting (CIL)

SUMMARY:
The aim of this multi-site randomized control trial will be is to assess the impact Systematic lighting on circadian rhythm entrainment, Inflammation, Neutropenic Fever and Symptom Burden among Multiple Myeloma Patients undergoing Autologous Stem Cell Transplantation. To achieve this aim, 200 multiple myeloma patients will receive one of two different light-treatments that are designed to promote circadian rhythm alignment. While receiving these light treatments, participants' sleep efficiency, urine melatonin levels, blood inflammatory cytokine levels and symptoms will be assessed over a 2-month period.

DETAILED DESCRIPTION:
Individuals undergoing Autologous Stem Cell Transplant (ASCT) experience major transplant-related complications including elevated symptom burden, high rates of neutropenic fever, and increases in inflammatory cytokines. These transplant-related complications are augmented by circadian rhythms disruption (CRD), which leads to misalignment between melatonin levels and sleep times. Since light is a strong synchronizer of circadian rhythms, the proposed multi-site randomized controlled trial (RCT) will investigate whether lighting designed to deliver circadian effective light that promotes circadian alignment, will: 1) promote higher nighttime melatonin levels and better nighttime sleep, 2) reduce pro-inflammatory cytokines, 3) lower rates of neutropenic fever and 4) improve symptom burden in cancer patients undergoing Autologous Stem Cell Transplant.

Hospital rooms for patients undergoing inpatient Autologous Stem Cell Transplant at the Mount Sinai Medical Center (MSMC) and at the Memorial Sloan Kettering Cancer Center (MSKCC)) will be retrofitted to install 1 of 2 lighting interventions, either circadian-effective (intervention) and circadian-ineffective (comparison) ambient light that may improve sleep.

1-2 weeks and no more than 2 months prior to transplant, participants will be given an Actiwatch, Daysimeter (personal light meter), sleep logs, questionnaires, and a urine collection kit to assess melatonin. One blood sample for cytokine analyses will be collected during one of the hospital visits prior to transplant. Blood draws are always done in the morning and always at a similar time for the same individual. The same outcomes (questionnaires, Actiwatch, Daysimeter, urine samples, blood samples) will be collected during transplant period and once, four weeks after engraftment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma diagnosis
* Scheduled to undergo their first Autologous Stem Cell Transplant procedure.
* 21years or older
* Able to provide informed consent.
* English-language proficient

Exclusion Criteria:

* Previous Autologous Stem Cell Transplant procedure
* Pregnancy
* Eye diseases which limit the ability of light to be processed
* Secondary cancer diagnosis within the last 5 years
* Severe sleep disorders
* History of bipolar disorder or manic episodes
* Severe psychological impairment
* Previous use of light therapy
* Active infection including COVID-19 infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Urinary Melatonin | Baseline visit and 3 days after the Autologous Stem Cell Transplant
  Participants will be given vials for collection and detailed instructions to void their bladders on AM rising and any prior nighttime voids starting 2 h prior to their normal bedtimes, at which time they will be asked to dim the lights down to a minimum and avoid using their self-luminous displays. Participants (and nurses) will collect each void during that overnight in a separate vial and to record the times of each voiding. Urinary melatonin-sulfate (6 sulfatoxymelatonin, aMT6s) measurements will be assayed using a commercially available ELISA kit (IBL International, Hamburg, Germany).

SECONDARY OUTCOMES:
Sleep Efficiency using Actigraphy at 7 days post-transplant | at 7 days post-transplant
  The participant will be asked to wear a wrist actigraph to monitoring sleep and activity, daily for 5 consecutive days. From the actigraphy data, change in sleep efficiency will be calculated. A higher sleep efficiency indicates improved sleep.
Sleep Efficiency using Actigraphy at 3 days after engraftment | at 3 days after engraftment
  The participant will be asked to wear a wrist actigraph to monitoring sleep and activity, daily for 5 consecutive days. From the actigraphy data, change in sleep efficiency will be calculated. A higher sleep efficiency indicates improved sleep.
Sleep Efficiency using Actigraphy at 4 weeks after engraftment | at 4 weeks after engraftment
  The participant will be asked to wear a wrist actigraph to monitoring sleep and activity, daily for 5 consecutive days. From the actigraphy data, change in sleep efficiency will be calculated. A higher sleep efficiency indicates improved sleep.
Inflammatory cytokine CRP levels at Baseline | At baseline, or during the hospital visit prior to transplant
  A blood sample will be drawn to measure Inflammatory cytokine CRP levels. A decrease in CRP levels indicates reduced inflammation.
Inflammatory cytokine CRP levels at 7 days following transplant | at 7 days following transplant
  A blood sample will be drawn to measure Inflammatory cytokine CRP levels. A decrease in CRP levels indicates reduced inflammation.
Inflammatory cytokine CRP levels at 3 days following engraftment | at 3 days following engraftment
  A blood sample will be drawn to measure Inflammatory cytokine CRP levels. A decrease in CRP levels indicates reduced inflammation.
Inflammatory cytokine CRP levels at 4 weeks following engraftment | at 4 weeks following engraftment
  A blood sample will be drawn to measure Inflammatory cytokine CRP levels. A decrease in CRP levels indicates reduced inflammation.
Number of Neutropenic Fevers at 7 days post-transplant | at 7 days post-transplant
  Physician notes on patient neutropenic fever will be obtained from medical records. Neutropenic fever will be defined as temperature of 38.2 C or higher and an absolute neutrophil count of less than 500 cells/mm. Physician notes are reviewed, and the number of times neutropenic fever is reported for each participant is recorded.
Number of Neutropenic Fevers at 3 days after engraftment | at 3 days after engraftment
  Physician notes on patient neutropenic fever will be obtained from medical records. Neutropenic fever will be defined as temperature of 38.2 C or higher and an absolute neutrophil count of less than 500 cells/mm. Physician notes are reviewed, and the number of times neutropenic fever is reported for each participant is recorded.
Number of Neutropenic Fevers at 4 weeks after engraftment | at 4 weeks after engraftment
  Physician notes on patient neutropenic fever will be obtained from medical records. Neutropenic fever will be defined as temperature of 38.2 C or higher and an absolute neutrophil count of less than 500 cells/mm. Physician notes are reviewed, and the number of times neutropenic fever is reported for each participant is recorded.
Circadian Light levels measured with Daysimeter (light monitor) at 7 days post-transplant | at 7 days post-transplant
  Participants will be asked to wear Daysimeters as a pendant or a pin during all waking times during the intervention weeks. Light measurements from Daysimeters used as pendants or pins are the closest to light measurements at eye level. The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the intervention weeks.
Circadian Light levels measured with Daysimeter (light monitor) at 3 days after engraftment | at 3 days after engraftment
  Participants will be asked to wear Daysimeters as a pendant or a pin during all waking times during the intervention weeks. Light measurements from Daysimeters used as pendants or pins are the closest to light measurements at eye level. The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the intervention weeks.
Circadian Light levels measured with Daysimeter (light monitor) at 4 weeks after engraftment | at 4 weeks after engraftment
  Participants will be asked to wear Daysimeters as a pendant or a pin during all waking times during the intervention weeks. Light measurements from Daysimeters used as pendants or pins are the closest to light measurements at eye level. The Daysimeter will also be used to monitor the total amount of circadian light received by the participant during the intervention weeks.
MD Anderson Symptom Inventory Score-Multiple Myeloma (MDASI-MM) at Baseline | At baseline, or during the hospital visit prior to transplant
  MDASI-MM, with well-established reliability and validity, is 19-item measure of cancer-related symptom burden. It assesses 13 core symptoms common across cancer types and treatments (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness/tingling). In addition, 6 items assess symptom-related interference. All 19 items are rated with reference to "the last 24 hours" on a scale from 0 to 10 with anchors at the extreme ends of the scale (for symptom items, 0 = "Not Present" and 10 = "As Bad As You Can Imagine"; for interference items 0 = "Did Not Interfere" and 10 = "Interfered Completely. Higher scores indicate higher symptom interference. The MDASI-Multiple Myeloma (MM) is the MDASI plus 7 additional items assessing symptoms specific to patients with MM (constipation, muscle weakness, diarrhea, sore mouth/throat, rash, difficulty concentrating and bone aches).
MD Anderson Symptom Inventory Score-Multiple Myeloma (MDASI-MM) at 7 days following transplant | at 7 days following transplant
  MDASI-MM, with well-established reliability and validity, is 19-item measure of cancer-related symptom burden. It assesses 13 core symptoms common across cancer types and treatments (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness/tingling). In addition, 6 items assess symptom-related interference. All 19 items are rated with reference to "the last 24 hours" on a scale from 0 to 10 with anchors at the extreme ends of the scale (for symptom items, 0 = "Not Present" and 10 = "As Bad As You Can Imagine"; for interference items 0 = "Did Not Interfere" and 10 = "Interfered Completely. Higher scores indicate higher symptom interference. The MDASI-Multiple Myeloma (MM) is the MDASI plus 7 additional items assessing symptoms specific to patients with MM (constipation, muscle weakness, diarrhea, sore mouth/throat, rash, difficulty concentrating and bone aches).
MD Anderson Symptom Inventory Score-Multiple Myeloma (MDASI-MM) at 3 days following engraftment | at 3 days following engraftment
  MDASI-MM, with well-established reliability and validity, is 19-item measure of cancer-related symptom burden. It assesses 13 core symptoms common across cancer types and treatments (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness/tingling). In addition, 6 items assess symptom-related interference. All 19 items are rated with reference to "the last 24 hours" on a scale from 0 to 10 with anchors at the extreme ends of the scale (for symptom items, 0 = "Not Present" and 10 = "As Bad As You Can Imagine"; for interference items 0 = "Did Not Interfere" and 10 = "Interfered Completely. Higher scores indicate higher symptom interference. The MDASI-Multiple Myeloma (MM) is the MDASI plus 7 additional items assessing symptoms specific to patients with MM (constipation, muscle weakness, diarrhea, sore mouth/throat, rash, difficulty concentrating and bone aches).
MD Anderson Symptom Inventory Score-Multiple Myeloma (MDASI-MM) at 4 weeks following engraftment | at 4 weeks following engraftment
  MDASI-MM, with well-established reliability and validity, is 19-item measure of cancer-related symptom burden. It assesses 13 core symptoms common across cancer types and treatments (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, lack of appetite, drowsiness, dry mouth, sadness, vomiting, and numbness/tingling). In addition, 6 items assess symptom-related interference. All 19 items are rated with reference to "the last 24 hours" on a scale from 0 to 10 with anchors at the extreme ends of the scale (for symptom items, 0 = "Not Present" and 10 = "As Bad As You Can Imagine"; for interference items 0 = "Did Not Interfere" and 10 = "Interfered Completely. Higher scores indicate higher symptom interference. The MDASI-Multiple Myeloma (MM) is the MDASI plus 7 additional items assessing symptoms specific to patients with MM (constipation, muscle weakness, diarrhea, sore mouth/throat, rash, difficulty concentrating and bone aches).
Perceived Stress Scale Score at Baseline | At baseline, or during the hospital visit prior to transplant
  Perceived Stress Scale is a 10-item self-report questionnaire that measures a person's self-reported evaluation of their perception of stressfulness in a situation over the past 1 month of their lives. It assesses a person's feelings and thoughts over a 1-month period. Participants rate each item on a 4-point scale (0 = "never," 1 = "almost never," 2 = "sometimes," 3 = "fairly often," 4 = "often") producing scores ranging from 0-40. Scores are obtained by reversing the scores on items 4,5,7 and 8 like so: 0=1,1=3,2=2,3=1,4=0, and then adding up the scores for each item to obtain a total score. Higher scores indicate greater stress.
Perceived Stress Scale Score at 7 days post-transplant | at 7 days post-transplant
  Perceived Stress Scale is a 10-item self-report questionnaire that measures a person's self-reported evaluation of their perception of stressfulness in a situation over the past 1 month of their lives. It assesses a person's feelings and thoughts over a 1-month period. Participants rate each item on a 4-point scale (0 = "never," 1 = "almost never," 2 = "sometimes," 3 = "fairly often," 4 = "often") producing scores ranging from 0-40. Scores are obtained by reversing the scores on items 4,5,7 and 8 like so: 0=1,1=3,2=2,3=1,4=0, and then adding up the scores for each item to obtain a total score. Higher scores indicate greater stress.
Perceived Stress Scale Score at 3 days following engraftment | at 3 days following engraftment
  Perceived Stress Scale is a 10-item self-report questionnaire that measures a person's self-reported evaluation of their perception of stressfulness in a situation over the past 1 month of their lives. It assesses a person's feelings and thoughts over a 1-month period. Participants rate each item on a 4-point scale (0 = "never," 1 = "almost never," 2 = "sometimes," 3 = "fairly often," 4 = "often") producing scores ranging from 0-40. Scores are obtained by reversing the scores on items 4,5,7 and 8 like so: 0=1,1=3,2=2,3=1,4=0, and then adding up the scores for each item to obtain a total score. Higher scores indicate greater stress.
Perceived Stress Scale Score at 4 weeks following engraftment | at 4 weeks following engraftment
  Perceived Stress Scale is a 10-item self-report questionnaire that measures a person's self-reported evaluation of their perception of stressfulness in a situation over the past 1 month of their lives. It assesses a person's feelings and thoughts over a 1-month period. Participants rate each item on a 4-point scale (0 = "never," 1 = "almost never," 2 = "sometimes," 3 = "fairly often," 4 = "often") producing scores ranging from 0-40. Scores are obtained by reversing the scores on items 4,5,7 and 8 like so: 0=1,1=3,2=2,3=1,4=0, and then adding up the scores for each item to obtain a total score. Higher scores indicate greater stress.
Patient-Reported Outcomes Measurement Information System -Sleep Disturbance Short Form (PROMIS-SD) Score at Baseline | At baseline, or during the hospital visit prior to transplant
  Participants will complete the 8-item PROMIS Sleep Disturbance Short Form (PROMIS-SD) during assessment periods to assess the pure domain of sleep disturbances among adults ages 18 and older. Participants rate each item on a 5-point scale (1 = "never," 2 = "rarely," 3 = "sometimes," 4 = "often," 5 = "always"), producing scores ranging from 8-40. Raw scores for the 8 items are summed for a global score; higher scores indicate greater severity of sleep disturbance.
Patient-Reported Outcomes Measurement Information System -Sleep Disturbance Short Form (PROMIS-SD) Score at 7 days post-engraftment | at 7 days following transplant
  Participants will complete the 8-item PROMIS Sleep Disturbance Short Form (PROMIS-SD) during assessment periods to assess the pure domain of sleep disturbances among adults ages 18 and older. Participants rate each item on a 5-point scale (1 = "never," 2 = "rarely," 3 = "sometimes," 4 = "often," 5 = "always"), producing scores ranging from 8-40. Raw scores for the 8 items are summed for a global score; higher scores indicate greater severity of sleep disturbance.
Patient-Reported Outcomes Measurement Information System -Sleep Disturbance Short Form (PROMIS-SD) Score at 3 days following engraftment | at 3 days following engraftment
  Participants will complete the 8-item PROMIS Sleep Disturbance Short Form (PROMIS-SD) during assessment periods to assess the pure domain of sleep disturbances among adults ages 18 and older. Participants rate each item on a 5-point scale (1 = "never," 2 = "rarely," 3 = "sometimes," 4 = "often," 5 = "always"), producing scores ranging from 8-40. Raw scores for the 8 items are summed for a global score; higher scores indicate greater severity of sleep disturbance.
Patient-Reported Outcomes Measurement Information System -Sleep Disturbance Short Form (PROMIS-SD) Score at 4 weeks following engraftment | at 4 weeks following engraftment
  Participants will complete the 8-item PROMIS Sleep Disturbance Short Form (PROMIS-SD) during assessment periods to assess the pure domain of sleep disturbances among adults ages 18 and older. Participants rate each item on a 5-point scale (1 = "never," 2 = "rarely," 3 = "sometimes," 4 = "often," 5 = "always"), producing scores ranging from 8-40. Raw scores for the 8 items are summed for a global score; higher scores indicate greater severity of sleep disturbance.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Fatigue Score at Baseline | At baseline, or during the hospital visit prior to transplant
  Participants, 18 years and older, will complete the 13-item PROMIS Fatigue Short Form items which asses a range of self-reported symptoms of fatigue from mild feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that decreases one's ability to execute daily activities and function normally in family or social roles. On the form, Participant Fatigue is divided by the impact of fatigue on physical, mental, and social activities. All items assess fatigue over the past 7 days. Participants will rate each item on a 5-point scale (1= "Not at all", 2= "A little bit", 3= "Somewhat", 4= "Quite a bit", 5= "Very much"). Scores will be summed to produce a total or raw score ranging from 8. (lowest score) to 40, with a higher score indicating more frequent fatigue. If all questions were responded to, a scoring table will be used to generate the T-score.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Fatigue Score at 7 days following transplant | at 7 days following transplant
  Participants, 18 years and older, will complete the 13-item PROMIS Fatigue Short Form items which asses a range of self-reported symptoms of fatigue from mild feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that decreases one's ability to execute daily activities and function normally in family or social roles. On the form, Participant Fatigue is divided by the impact of fatigue on physical, mental, and social activities. All items assess fatigue over the past 7 days. Participants will rate each item on a 5-point scale (1= "Not at all", 2= "A little bit", 3= "Somewhat", 4= "Quite a bit", 5= "Very much"). Scores will be summed to produce a total or raw score ranging from 8. (lowest score) to 40, with a higher score indicating more frequent fatigue. If all questions were responded to, a scoring table will be used to generate the T-score.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Fatigue Score at 3 days following engraftment | at 3 days following engraftment
  Participants, 18 years and older, will complete the 13-item PROMIS Fatigue Short Form items which asses a range of self-reported symptoms of fatigue from mild feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that decreases one's ability to execute daily activities and function normally in family or social roles. On the form, Participant Fatigue is divided by the impact of fatigue on physical, mental, and social activities. All items assess fatigue over the past 7 days. Participants will rate each item on a 5-point scale (1= "Not at all", 2= "A little bit", 3= "Somewhat", 4= "Quite a bit", 5= "Very much"). Scores will be summed to produce a total or raw score ranging from 8. (lowest score) to 40, with a higher score indicating more frequent fatigue. If all questions were responded to, a scoring table will be used to generate the T-score.
Patient-Reported Outcomes Measurement Information System (PROMIS)- Fatigue Score at 4 weeks following engraftment | at 4 weeks following engraftment
  Participants, 18 years and older, will complete the 13-item PROMIS Fatigue Short Form items which asses a range of self-reported symptoms of fatigue from mild feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that decreases one's ability to execute daily activities and function normally in family or social roles. On the form, Participant Fatigue is divided by the impact of fatigue on physical, mental, and social activities. All items assess fatigue over the past 7 days. Participants will rate each item on a 5-point scale (1= "Not at all", 2= "A little bit", 3= "Somewhat", 4= "Quite a bit", 5= "Very much"). Scores will be summed to produce a total or raw score ranging from 8. (lowest score) to 40, with a higher score indicating more frequent fatigue. If all questions were responded to, a scoring table will be used to generate the T-score.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn Schoool of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
Analyzed data from the study will be shared, as this information is more relevant to the research. IDP does not need to be shared for this research.